CLINICAL TRIAL: NCT05132283
Title: Image-guided Lymphadenectomy Within Urologic Regions of Interest in AMIGO
Brief Title: Urologic Lymphadenectomy in AMIGO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Matthew Mossanen, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-372
Record Dates: First submitted 2021-11-01; First posted 2021-11-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Urologic Cancer; Lymph Node Metastasis
Keywords: Urologic Cancer; Lymph Node Metastasis
MeSH Terms: conditions — Urologic Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Urologic Lymphadenectomy in AMIGO (Experimental): Participants will undergo Lymphadenectomy per standard of care with the navigation systems (3D Slicer and Monaco) used to locate the abnormal lymph node(s).
  Interventions: Device: 3D Slicer; Device: Monaco

INTERVENTIONS:
Device: 3D Slicer — Navigational device used during surgery to locate abnormal lymph nodes.
Device: Monaco — Navigational device used during surgery to locate abnormal lymph nodes.

SUMMARY:
This research study involves the use of two navigation systems, the 3D Slicer-based navigation system, and the Siemens Monaco systems, to simplify the complexity of image-guided lymphadenectomy procedures (surgery to remove one or more lymph nodes) in patients with urological cancer.

DETAILED DESCRIPTION:
This research study involves the use of two navigation systems, the 3D Slicer-based navigation system, and the Siemens Monaco systems, which will simplify the complexity of image-guided lymphadenectomy procedures (surgery to remove one or more lymph nodes).

The U.S. Food and Drug Administration (FDA) has not approved the navigation systems (3D Slicer and Monaco) as a treatment for any disease.

In this research study, our hypothesis is that the use of the navigation systems (3D Slicer and the Siemens Monaco system) may simplify the complexity of laparoscopic lymphadenectomy (The procedure in which a small incision is made in the lower abdomen to reach the lymph nodes) in regions of urologic interest, by resulting in better visualization and more accurate localization of the diseased lymph node and allowing for improved surgical and patient outcomes, fewer complications, and better clinician performance.

The long-term goal of our program is to demonstrate that the navigation system (3D Slicer and the Siemens Monaco system) increase the efficiency and reduce the morbidity or the likelihood of any medical problems associated with the resection or removal of radiologically defined lesions, within urologic regions of interest, associated with any type of urologic cancer. The first clinical application of the system will be in resecting radiologically positive lymph nodes displayed by CT or FDG PET (an imaging test used to identify lymphomas and other cancers) in the Advanced Multimodality Image-Guided Operating (AMIGO) Suite at Brigham and Women's Hospital (BWH).

The navigation system has been used with similar protocols, specifically 5 parathyroid surgeries, 13 tracked endoscopic ultrasound (minimally invasive procedure to assess digestive and lung diseases) and over 30 tracked colonoscopy experiments (exam used to detect changes or abnormalities in the large intestine (colon) and rectum) on human subjects at BWH with no difficulties or reportable incidents.

It will take you up to 4 weeks to complete this study. During that time you will have two study visits and one standard of care follow-up visit.

The research study procedures include: screening for eligibility and study treatment including evaluations and standard of care follow-up visits.

It is expected that about 20 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent before any trial-related procedure is undertaken that is not part of the standard patient management
* Subjects aged ≥ 18 years. Selected patients must have a confirmed or suspected diagnosis of disease in urologic regions of interest, with scheduled confirmatory surgical biopsy.
* Subjects must have had a CT, PET or MR examination of acceptable quality at Brigham and Women's Hospital within the prior month.
* Subjects must also be scheduled to undergo lymphadenectomy for a urologic cancer within the following urologic regions of interest: Bladder, Prostate, Testicular, Kidney, Urethral, and Penile.
* Subjects must also be scheduled to undergo a laparoscopic lymphadenectomy within the AMIGO OR

Exclusion Criteria:

* Severely impaired renal function with an EGFR < 30 mL/min/body surface area
* Evidence of any significant, uncontrolled comorbid condition that could affect compliance with the protocol or interpretation of the results, which is to be judged at the discretion of the PI
* History of hypersensitivity or other contraindication to contrast media
* Contraindication to general anesthesia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-08-26 (Estimated); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Completing Intended Procedure (Feasibility) | One month, up to 45 days after registration
  The Slicer-Monaco prototype navigation platform will be used to resect enlarged and/or fluorodeoxyglucose avid lymph nodes. The successful navigational use of this platform will be considered as completed. The proportion of patients completing this intended procedure will be reported.

SECONDARY OUTCOMES:
Proportion of Patients with Laparoscopic Videos Recorded | One month, up to 45 days from registration
  During the first phase of the project on 10 patients, we will store real-time laparoscopic videos using the KARL STORZ 3D Video system that can be analyzed offline. During the second phase of 10 patients, we will provide an optional video overlay option in the navigation system. The navigation system will be similar to that used on the first 10 patients. The only difference will be that the virtual endoscopy view will be overlaid on the laparoscopy video in the 3D Slicer navigation system.
Path length Kinematic Metric | One month, up to 45 days after registration
  The kinematic metric of path length will be computed using recorded data from the navigation system. Mean path length scores for all patients will be reported for each kinematic measure.
Velocity Kinematic Metric | One month, up to 45 days after registration
  The kinematic metric of velocity will be computed using recorded data from the navigation system. Mean velocity scores for all patients will be reported for each kinematic measure.
Acceleration Kinematic Metric | One month, up to 45 days after registration
  The kinematic metric of acceleration will be computed using recorded data from the navigation system. Mean acceleration scores for all patients will be reported for each kinematic measure.
Jerk Kinematic Metric | One month, up to 45 days after registration
  The kinematic metric of jerk will be computed using recorded data from the navigation system. Mean jerk scores for all patients will be reported for each kinematic measure.
Mental/Physical/Temporal Demand on Physician | One month, up to 45 days after registration
  The mental, physical and temporal demand on physicians will be assessed using the NASA Task Load Index (NASA-TLX), a multidimensional assessment tool that rates perceived workload in order to assess the performance of a task. The NASA task load index has a scoring range of 1 to 10 for mental demand, physical demand, temporal demand, effort, and frustration with 1 representing a very low value and 10 representing a very high value. A mean score out of 10 will be given for each operation and a mean score for all 20 operations will be given (out of 10). Assessment will be filled out by investigators.
Mean absolute difference in distance from Instruments to Organs | One month, up to 45 days after registration
  The accuracy of localization of the organs will be quantified by pointing to specific structures and evaluating the distance of the registered instrument from the structures in the image space.
Further, the pathology of the lymph node resected using the navigation system will be compared to the other lymph nodes resected in urologic regions of interest. | One month, up to 45 days after registration
  To ensure quality control of the procedure, the lymph node removed with the navigation system will be compared to the other lymph nodes resected in urologic regions of interest without the use of the navigation system.
  The unit of measure will be the accuracy of targeting the PET-avid lymph node as confirmed by pathology, i.e., binary decision variable for two categories (using the navigation system or not). Using the navigation system: malignant or not, versus not using with the navigation system: malignant or not. The measurement tool will be the pathological analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Mossanen, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation